CLINICAL TRIAL: NCT00024518
Title: Ingested Interferon-Alpha: Prolongation or Permanence of the "Honeymoon" Phase in Newly Diagnosed Diabetes Mellitus
Brief Title: Interferon-Alpha for Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010249; 01-DK-0249
Record Dates: First submitted 2001-09-19; First posted 2001-09-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Insulin-Dependent Diabetes Mellitus
Keywords: Diabetes; Immunotherapy; Study Drug; Insulin Dependent Diabetes; Diabetes Mellitus; TIBM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): placebo was prepared as saline alone with 6mg human serum albumin (HSA). Subjects orally ingested one vial each morning before breakfast with at least 150mL water.
  Interventions: Other: Placebo
- 5,000 Units hrIFN-alpha (Experimental): hrIFN-alpha = human recombinant interferon-alpha. 5,000 units was prepared along with saline and 6mg HSA. Subjects orally ingested one vial each morning before breakfast with at least 150mL water.
  Interventions: Drug: 5,000 hrINF-alpha
- 30,000 hrIFN-alpha (Experimental): 30,000 units hrIFN-alpha was prepared along with saline and 6mg HSA. Subjects orally ingested one vial each morning before breakfast with at least 150mL water.
  Interventions: Drug: 30,000 units hrINF-alpha

INTERVENTIONS:
Drug: 30,000 units hrINF-alpha
  Other Names: Human Recombinant Interferon-alpha
  Arms: 30,000 hrIFN-alpha
Drug: 5,000 hrINF-alpha
  Other Names: Human Recombinant Interferon-alpha
  Arms: 5,000 Units hrIFN-alpha
Other: Placebo — placebo was prepared as saline alone with 6mg human serum albumin (HSA).
  Arms: Placebo

SUMMARY:
This study will see if interferon-alpha given early in the disease can stop or slow the immune attack on insulin-producing cells. In addition, the study will examine the safety and efficacy of interferon-alpha (given by mouth) to protect beta cell function. Patients between 3 and 25 years of age with Type 1 Diabetes Mellitus less then six weeks may be eligible for this study. All study-related tests and medications at the NIH Clinical Center are provided at no cost.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) results from autoimmune destruction of the insulin-producing pancreatic beta-cells. The onset of clinical symptoms represents the endpoint of a chronic progressive decline in beta-cell function when the number of functional beta-cells descends below the critical mass required for maintenance of euglycemia ([1], [2]). However, the pancreas still retains the ability to produce a substantial amount of insulin. The goal of secondary prevention in T1DM is to avert further destruction of the remaining beta-cells and therefore delay or stop entry into the final stages of the disease associated with end organ damage.

The rationale for this study is to interfere with the autoimmune beta-cell destruction early on in order to preserve as much residual endogenous insulin production as possible. We plan to administer oral interferon-alpha (IFN-a) on a daily basis, which has been shown to modify the clinical course of diabetes, to alter cytokine release, and reduce expression of T cell activation markers in an animal model ([3]) and a pilot project in humans (S. Brod, University of Texas, unpublished data). The one-year study is designed as a double blind randomized protocol using either 5,000 or 30,000 units of IFN-a versus placebo. Five centers will participate in this protocol (University of Texas Health Science Center in Houston; Dallas; Children's Hospital, St. Paul, MN; Kansas City and NIH, Bethesda, Maryland).

ELIGIBILITY:
* INCLUSION CRITERIA:

T1DM of less than 6 weeks duration in patients between 3 and 25 years of age.

Besides T1DM, no concurrent illness.

EXCLUSION CRITERIA:

Treatment with immunosuppressive or immunostimulatory medications such as azathioprine, nicotinamide, superoxide dismutase-desferroxamine, aminoguanidine, oral insulin or other experimental therapies at the present time or in the past.

Abnormal pre-treatment white blood cell count (WBC) or thrombocytopenia.

Known active diseases, e.g. cardiac, renal, hepatic diseases or immunodeficiency.

History of cancer, neuropathy seizure disorders (except typical history of febrile seizures in childhood), peripheral vascular disease, coagulation abnormalities, autoimmune disease (except type 1 diabetes) or cerebrovascular disease.

Ongoing use of medications known to influence glucose tolerance (e.g. sulfonylureas, metformin, diphenylhydantoin, thiazide or other potassium depleting diuretics, beta-adrenergic blockers, niacin) except insulin.

Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Inability to give informed consent or assent.

Participation in a clinical trial within the previous 6 weeks.

Lactating or pregnant female individual (individuals will be advised not to volunteer for the protocol if they plan to become pregnant during the time of the study and they are instructed to use an effective method of contraception).

Age above 25 years, since there may be several subtypes of T1DM.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2001-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
C-Peptide Level | Baseline - 3mth, 6mnth, 9mnth, 12mnth
  The Connecting Peptide, or C-peptide, is a short 31-amino-acid protein that connects insulin's A-chain to its B-chain in the proinsulin molecule.

SECONDARY OUTCOMES:
Serum glucose | baseline - 3mths, 6mnths, 9mnths, 12mnths
  Serum glucose or blood sugar measurements determine how much sugar is in the blood.
Hemoglobin A1C | Baseline - 3mnths, 6mnths, 9mnths, 12mnths
  a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina I Rother, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Staley A Brod, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (5):
- United States (5):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Children's Hospital - St. Paul, Saint Paul, Minnesota
  - Children's Hospital - Kansas City, Kansas City, Missouri
  - University of Texas, Dallas, Dallas, Texas
  - University of Texas, Houston, Houston, Texas

REFERENCES:
- [Background] Atkinson MA, Maclaren NK. The pathogenesis of insulin-dependent diabetes mellitus. N Engl J Med. 1994 Nov 24;331(21):1428-36. doi: 10.1056/NEJM199411243312107. No abstract available. PMID 7969282
- [Background] Eisenbarth GS. Type I diabetes mellitus. A chronic autoimmune disease. N Engl J Med. 1986 May 22;314(21):1360-8. doi: 10.1056/NEJM198605223142106. No abstract available. PMID 3517648
- [Background] Brod SA, Malone M, Darcan S, Papolla M, Nelson L. Ingested interferon alpha suppresses type I diabetes in non-obese diabetic mice. Diabetologia. 1998 Oct;41(10):1227-32. doi: 10.1007/s001250051056. PMID 9794112
- [Result] Rother KI, Brown RJ, Morales MM, Wright E, Duan Z, Campbell C, Hardin DS, Popovic J, McEvoy RC, Harlan DM, Orlander PR, Brod SA. Effect of ingested interferon-alpha on beta-cell function in children with new-onset type 1 diabetes. Diabetes Care. 2009 Jul;32(7):1250-5. doi: 10.2337/dc08-2029. PMID 19564474
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DK-0249.html